CLINICAL TRIAL: NCT01944319
Title: Clinical Evaluation of a Meropenem Dosage Strategy Based on a Population Pharmacokinetic-pharmacodynamic Model in Lower Respiratory Tract Infection Patients
Brief Title: Meropenem Dosage Strategy Based on PPK Model
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Qingtao Zhou (Other)
Responsible Party: Sponsor-Investigator, Qingtao Zhou, Associate professor, Peking University Third Hospital
Organization: Peking University Third Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 75505-01
Record Dates: First submitted 2013-07-02; First posted 2013-09-17 (Estimated); Results first posted 2016-02-25 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2016-01

CONDITIONS: Lower Respiratory Tract Infection
Keywords: Infection; Meropenem; Pharmacokinetics; Pharmacodynamics
MeSH Terms: conditions — Infections | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group (Active Comparator): The participants in control group will accept routine meropenem therapy
  Interventions: Drug: Routine meropenem therapy
- Study group (Experimental): The participants in study group will accept meropenem therapy based on a PPK and PD model.
  Interventions: Drug: Meropenem therapy based on a PPK and PD model

INTERVENTIONS:
Drug: Routine meropenem therapy — Participants in control group will accept meropenem therapy with regimen routinely decided by attending physician
  Other Names: Standard care
  Arms: Control group
Drug: Meropenem therapy based on a PPK and PD model — Participants in study group will accept meropenem therapy based on a software developed from a PPK and PD model
  Other Names: Experimental meropenem therapy
  Arms: Study group

SUMMARY:
To evaluate the clinical and economical benefits of a meropenem dosage strategy based on a population pharmacokinetic(PPK)-pharmacodynamic(PD) model in lower respiratory tract infection patients.

DETAILED DESCRIPTION:
* Subjects:lower respiratory tract infection patients
* Study design:randomized control study.The patients in study group will accept meropenem therapy with the regimen decided by a software developed from a PPK-PD model. The patients in control group will accept meropenem therapy with the regimen decided by attending physician.
* Primary endpoint: clinical successful rate of meropenem therapy. The clinical efficiency of meropenem therapy will be evaluated one week later from stop of meropenem therapy.
* Second endpoint: amount of used antibiotics and bacteriological successful rate.

ELIGIBILITY:
Inclusion Criteria:

* Sixty years and older patients hospitalized at the Peking University Third Hospital with community-acquired or hospital-acquired lower respiratory tract infection.
* Bacilli was idolated from lower respiratory tract specimens within 48 hours prior to study enrollment.
* The pathogen was sensitive to meropenem.
* Received broad-spectrum antibiotic therapy less than 24 hours, or no improvement after antibiotic therapy and pathogen was resistant to the used antibiotics.

Exclusion Criteria:

* Had documented hypersensitivity to carbapenems.
* More than one pathogenic Gram-negative bacillus was isolated lower respiratory tract specimens.
* Positive HIV antibody titre.
* Had known or suspected tuberculosis or other infections caused by Gram-positive cocci, viruses or fungi at baseline.

Ages: 60 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2013-07; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Qingtao Zhou, M.D., Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospita, Haidian District, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhou QT, He B, Shen N, Liang Y, Sun LN. Meropenem Dosing Based on a Population Pharmacokinetic-Pharmacodynamic Model in Elderly Patients with Infection of the Lower Respiratory Tract. Drugs Aging. 2017 Feb;34(2):115-121. doi: 10.1007/s40266-016-0431-9. PMID 28097633

RESULTS

PARTICIPANT FLOW:
Groups:
- Control Group: Meropenem therapy with regimen routinely decided by attending physician
- Study Group: Patients in Study group will accept meropenem therapy based on PPK and PD parameter.
  Meropenem therapy based on PPK and PD: Meropenem therapy with regimen decided by a software developed from a PPK model and clinical PD parameter
Period: Overall Study
Arm/Group | Control Group | Study Group
Started | 40 | 39
Completed | 40 | 39
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Study Group | Total
Number analyzed (Participants) | 40 | 39 | 79
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 79 [74 to 87] | 78 [76 to 84] | 79 [76 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 10 | 26
  Male | 24 | 29 | 53
Region of Enrollment [Number; unit: participants]
  China | 40 | 39 | 79

OUTCOME MEASURES:

1. Primary Outcome: Clinical Success Rate
Description: The clinical success or failure of meropenem therapy will be evaluated one week after stop of antibiotic therapy.
  Clinical success was defined as cure or improvement of all signs and symptoms caused by the infection and no requirement for additional antibacterial therapy.
  Clinical failure was defined as a persistence or worsening of any new clinical sign or symptom, development of any new clinical signs or symptoms of infection, or the requirement for other systemic antimicrobial therapy at the end of meropenem therapy.
Time Frame: One week after antibiotic therapy finished.
Measure: Number; unit: participants
Groups:
- Study Group: The participants in stusy group will accept meropenem therapy based on a PPK and PD model.
Arm/Group | Control Group | Study Group
Number analyzed (Participants) | 40 | 39
participants | 28 | 35

2. Secondary Outcome: Amount of Used Antibiotics
Description: Record the amount of antibiotics usage during antibiotic therapy
Time Frame: participants will be followed for the duration of antibiotic therapy, an average of 10 days
Measure: Median (Inter-Quartile Range); unit: grams
Arm/Group | Control Group | Study Group
Number analyzed (Participants) | 40 | 39
grams | 19.0 [12.0 to 29.5] | 15.0 [7.5 to 24.0]

3. Secondary Outcome: Bacteriological Success Rate
Description: The bacterial success or failure will be evaluated at the end of meropenem therapy.
  Bacteriological success including eradication and presumed eradication. Bacteriological failure including persistence and presumed persistence.
Time Frame: At the end of meropenem therapy, an average of 10 days.
Measure: Number; unit: participants
Arm/Group | Control Group | Study Group
Number analyzed (Participants) | 40 | 39
participants | 24 | 28

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Control Group | Study Group
Serious Adverse Events (participants affected / at risk) | 4/40 | 0/39
Other Adverse Events (participants affected / at risk) | 0/40 | 0/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Group (N=40) | Study Group (N=39)
Death (Vascular disorders) | 4 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes